CLINICAL TRIAL: NCT00119418
Title: TU 025 Keishi Bukuryo Gan for Post-Menopausal Hot Flash Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Plotnikoff, Gregory A., M.D. (Individual)
Collaborators: Tsumura and Company, Tokyo, Japan (Industry); University of Minnesota (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0402M56292; M01-RR00400 NIH; M01RR000400 (NIH)
Record Dates: First submitted 2005-07-04; First posted 2005-07-13 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2005-07

CONDITIONS: Hot Flashes; Menopause
Keywords: hot flash; menopause; herbal medicine; kampo; alternative medicine
MeSH Terms: conditions — Hot Flashes

INTERVENTIONS:
Drug: TU 025 Keishi Bukuryo Gan

SUMMARY:
This study tests to see if TU 025 Keishi Bukuryo Gan reduces the frequency and severity of hot flashes in post-menopausal American women. This study will also estimate the best dose amount and determine the common short-term side effects and risks.

DETAILED DESCRIPTION:
Menopause is a natural transition in a woman's hormonal state associated with the cessation of ovulation and menstruation. For approximately 80% of peri-menopausal women, menopause may be defined by the experience of uncomfortable symptoms such as hot flashes, night sweats, dyspareunia, urinary frequency, sleep disturbance, fatigue, depression and anxiety.

Hot flashes are the most common complaint of perimenopausal and postmenopausal Western women. Approximately 10-20% of postmenopausal women find such symptoms nearly intolerable. Nearly one-third of postmenopausal women experience disruptive hot flashes for 5 years after natural menopause and approximately 20% experience hot flashes for 15 years.

Menopause has been understood as an estrogen deficiency state from which women are placed at great risk for osteoporosis, colon cancer and heart disease. For symptom management, as well as for disease prevention, the medical response for 20 years has been hormone replacement therapy (HRT). In recent years, as many as 38% of US women between ages 50 and 74 years were using HRT.

For menopause hormone therapy, in 2005, counseling patients from an evidence-based perspective means informing patients of the significantly increased risk of dementia, breast cancer,endometrial cancer,venous thromboembolism and gallbladder disease. Additionally, physicians must also state that hormone therapy increases the risk of cardiovascular events (heart attack or strokes) in women with or without pre-existing heart disease. Furthermore, well-done studies demonstrate that hormone therapy does not enhance health-related quality of life.

For this reason, there is great interest in non-hormonal alternatives for menopausal hot flash management. The current standard of care, based on controlled clinical trials in women with breast cancer, is the use of SSRI anti-depressants such as venlafaxine. However, many women seek other options.

In Japan, TJ25 Keishi Bukuryo Gan is a leading non-hormonal prescription agent for management of menopausal hot flashes. However, no clinical data exists on its effectiveness in American women.

This is a pilot phase II clinical study to estimate the effectiveness of TU-25 Keishi Bukuryo Gan for reduction of both the severity and the frequency of hot flashes in healthy postmenopausal American women. This study will also estimate the best dose and determine the common short-term side effects and risks.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged 45-58 with an adequate hot flash frequency severity score. Post-menopause is defined as amenorrhea for at least 12 months, or post-hysterectomy for more than one year with follicle-stimulating hormone levels greater than or equal to 40 mIU/mL and estradiol (E2) levels of less than or equal to 20 pg/mL, or greater than two months post oophorectomy.
* All subjects must be up to date with both pap and mammogram screening by the US Preventative Services Taskforce Guidelines for the length of the trial.
* All subjects on any prescription medication need the approval of their prescribing physician for participation in the trial.

Exclusion Criteria:

* Concurrent hot flash therapies (prescription medications including hormones, antidepressants, SERMs, gabapentin or over the counter supplements)
* Moderately severe disease state(s) or diseases that affect absorption/metabolism, or diseases that mimic menopausal hot flashes.
* Inability to swallow vitamin size pills
* Beck depression inventory score greater than 11
* Greater than 10 cigarettes per day
* Abnormal liver function
* Treated or untreated hypertension greater than 160/90.
* BMI greater than 36
* Inability to give consent or commit to the length of the trial
* Known hypersensitivity to ingredients
* Physician judgment

Ages: 45 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2004-11; Study Completion 2006-02

PRIMARY OUTCOMES:
frequency and severity of hot flashes by Mayo Hot Flash Diary

SECONDARY OUTCOMES:
sleep quality by the Pittsburgh Questionnaire
bodyweight/BMI by standard measurements
quality of menopausal life by Greene Climacteric Scale
lipid profile by laboratory test
liver function profile by laboratory test
hormone profile by laboratory test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota General Clinical Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Plotnikoff GA, Watanabe K, Torkelson C, La Valleur J, Radosevich DM. The TU-025 keishibukuryogan clinical trial for hot flash management in postmenopausal women: results and lessons for future research. Menopause. 2011 Aug;18(8):886-92. doi: 10.1097/gme.0b013e31821643d9. PMID 21738077